CLINICAL TRIAL: NCT05395754
Title: Assessing the Feasibility and Preliminary Impact of a mHealth App on Reducing STI Risk in Black MSM PrEP Users
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Principal Investigator, Meredith Clement, Assistant Professor, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2268
Record Dates: First submitted 2022-01-14; First posted 2022-05-27 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: STI; Sexually Transmitted Diseases; Pre-exposure Prophylaxis
Keywords: BMSM; STI; Sexually Transmitted Infection; Mobile health; PrEP; pre-exposure prophylaxis; MSM
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCheck (Experimental): Participants allocated to the intervention arm will receive the intervention (use of the PCheck app) for 12 months of follow-up. Participants will be encouraged to use the app as much as they wish throughout the study and will be informed that there will be no set expectation for how frequently they must use the app, although they will be encouraged to use it regularly to "thoroughly test it". The app will send notification reminders to "check in" (in other words, use the daily check-in feature to track their mood, stress, and behaviors related to STI-prevention over time). The notification settings can be adjusted in phone settings by the participant. To encourage peer support and a sense of community, users can interact with community members anonymously through a message board, monitored by research staff. Participants in the intervention will continue routine PrEP care and STI testing through the clinic.
  Interventions: Device: App Intervention
- Routine Care (No Intervention): Participants in the routine care arm will continue routine PrEP care and STI testing through the clinic.

INTERVENTIONS:
Device: App Intervention — Use of the PCheck app, an app encouraging STI prevention behaviors.
  Arms: PCheck

SUMMARY:
The study will recruit 120 Black men who have sex with men (BMSM) from the local area, New Orleans. The main purpose of this research study is to test the effect of a new smartphone application, "PCheck," on reducing the incidence of STIs, compared to routine care through the LSU-Crescent Care Sexual Health/PrEP Clinic.

DETAILED DESCRIPTION:
This unblinded, randomized study will determine the feasibility and preliminary impact of our adapted PCheck app in reducing STI infections in Black MSM PrEP users. Over 24 months, the research staff will prospectively enroll BMSM entering or already engaged in PrEP care. Participants will be randomly allocated 2:1 to the PCheck intervention versus standard of care using an automated system for randomization; the rationale for heavier allocation to the intervention is to allow for more participants to interact on the app (colleagues at the University of Virginia who have tested a similar app advised that a "critical mass" of roughly 20 participants using the community forum is needed for discussions to begin organically). Randomization will occur upon first meeting with the clinical research coordinator (CRC).

At enrollment, those randomized to the intervention arm will receive hands-on app onboarding training by the CRC. The training is anticipated to take 15-30 minutes and will include an overview of the app's features and how to use each, coaching about using the daily check-in feature to record mood, stress levels, and recent sexual activity and condom use, guidance on creating an anonymous introductory post to the community board, and practice using each of the PCheck features. Participants allocated to the intervention arm will receive the intervention (use of the PCheck app) for 24 months of follow-up. Participants will be encouraged to use the app as much as they wish throughout the study and will be informed that there will be no set expectation for how frequently they must use the app, although they will be encouraged to use it regularly to "thoroughly test it". The app will send notification reminders to "check in" (in other words, use the daily check-in feature to track their mood, stress, and behaviors related to STI-prevention over time). The notification settings can be adjusted in phone settings by the participant.

For participants receiving the app intervention, study staff will also schedule a follow-up call within two weeks after enrollment to encourage engagement, to talk through any difficulties that arise with using the app and to troubleshoot. During the 24 months of enrollment, study staff will contact participants at the 1, 2, 4, and 12 week marks after they stop showing usage on the app to encourage re-engagement and address any technical or other barriers.

To encourage engagement with the app, the research team will post short quizzes on the app's landing page and reminders about them on the community message board. The study will pilot once-a-day trivia questions, and adjust the frequency of trivia postings pending on participant engagement and/or feedback. Each set of trivia questions will take a couple minutes to complete and will ask 1-2 questions such as general knowledge about STIs, sexual health and wellness, and/or general New Orleans-specific or LGBTQI+ history. All participants who complete four of the quizzes for the week will be entered into a raffle for an additional $10 loaded onto their Clincard.

For app users, data will be extracted directly from the PCheck app, including app usage and data from the app's check-in, PrEP adherence, and STI prevention features. App data will be de-identified except for anonymous username and study ID number, which can be linked to identifying information in order to contact individuals not showing usage on the app, as described above.

For all participants, STI (syphilis, gonorrhea, chlamydia, HIV) screening will occur every three months and HCV screening every 6-12 months over 24 months of follow-up as part of routine care. Every three months, all participants will also complete self-administered questionnaires with demographic, social, and behavioral assessments. Participants allocated to the standard of care control group will be informed that their participation entails attending routine PrEP appointments, including STI screening, and completing the quarterly surveys. For those in the intervention arm, participants will also answer questions aimed at assessing app acceptability, feasibility, and usability.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender man who has sex with cisgender men (MSM) including gay, bisexual, or other MSM
* Age 18-35 years
* Black race or multi-racial including Black race
* Prescribed, administered or otherwise taking PrEP via routine care or PrEP clinical trial
* Smartphone possession

Exclusion criteria:

* Unable to read and write
* Not fluent in English

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
STI incidence | 24 months
  New diagnosis of syphilis, gonorrhea, chlamydia, or hepatitis C per 100 person-years. Number of new HIV diagnoses.

SECONDARY OUTCOMES:
Social Support | 24 months
  Scaled score on the Social Provisions Scale-10. The minimum score is 10 and maximum score is 40. Higher scores indicate a higher degree of social support.
Social Isolation | 24 months
  Scaled score on the Patient-Reported Outcomes Measurement Information System (PROMIS) Social Isolation Subscale. Higher scores indicate a higher degree of social isolation or disconnection from others. The minimum score is 4 and maximum score is 20.

CONTACTS AND LOCATIONS:
Overall Officials: Meredith Clement, MD, Principal Investigator — LSUHSC
Locations (2):
- United States (2):
  - CrescentCare PrEP Clinic, New Orleans, Louisiana
  - LSU-CrescentCare Sexual Health Center, New Orleans, Louisiana

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/54/NCT05395754/ICF_000.pdf